CLINICAL TRIAL: NCT00427102
Title: A Phase 1 Study of Oral MRX-1024 in Combination With Standard Fractionation Radiation Therapy and High-Dose Cisplatin in Patients With Squamous Cell Carcinoma of the Head and Neck Following Surgical Resection
Brief Title: MRX, Radiation, and Chemotherapy for Patients With Resected Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No subjects enrolled and PI went to another facility
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J-0657; 06-01
Record Dates: First submitted 2007-01-24; First posted 2007-01-26 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer; Resected Head and Neck Cancer; Mucositis
Keywords: Oral MRX-1024; High-Dose Cisplatin Chemotherapy; Standard Radiation Therapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Mucositis

INTERVENTIONS:
Drug: Oral MRX-1024
Procedure: Standard Fractionation Radiation Therapy
Drug: High-Dose Cisplatin Chemotherapy

SUMMARY:
Rationale for Study

Oral mucositis is a major complication arising from contemporary chemoradiation treatment of patients with head and neck cancer.

No effective therapy exists to prevent this complication in this population. MRX-1024 is an investigational agent that has demonstrated in in vitro and in vivo experiments to have the potential to exert a protective effect in normal mucosa cells, without interfering with the intended antitumor effect of radiation.

A pilot Phase 1 study of MRX-1024 was conducted in India in patients with head and neck cancer receiving radiation alone or radiation in combination with cisplatin or carboplatin. MRX 1024 doses of 100 mgkg given orally twice a day, five days a week during radiation treatment cycles, were well tolerated and appeared to exert a protective effect against the development of severe mucositis.

Twice daily doses of MRX 1024 impose a certain level of inconvenience to the patient, to their clinic companion, and to the general work flow within radiation oncology clinics.

This study is designed to study the safety and pharmacokinetics of both single daily dose and twice daily dose regimens of oral MRX 1024 given in conjunction with daily radiation fractions and intermittent high-dose cisplatin to patients with high-risk for recurrence head and neck cancer following surgical resection. The study will also document the incidence and severity of oral mucositis that occurs following such therapy. The results will be instrumental in determining the regimen of MRX 1024 to use in subsequent definitive clinical trials.

DETAILED DESCRIPTION:
TREATMENT PLAN

Study Phases

Each patient progresses through five study phases.

MRX 1024 Cohorts, Dose Levels and Treatment

Five successive dose levels are planned.

MRX 1024 Combination Treatment Phase Cohort Combination Treatment Phase MRX 1024 Schedule

MRX 1024 Dose Level once daily in cohorts 1, 2, and 3 twice daily in cohorts 4 and 5)

Initial Cohort Size 1 One daily dose given 30 minutes before each dose of RT 50 mg kg 3 patients 2 One daily dose given 30 minutes before each dose of RT 75 mg kg 3 patients 3 One daily dose given 30 minutes before each dose of RT 100 mg kg 3 patients 4a Two daily doses: one given 30 minutes before and one given 30 minutes after each dose of RT 75 mg kg 3 patients 5a Two daily doses: one given 30 minutes before and one given 30 minutes after each dose of RT 100 mg kg 3 patients

Because of the logistics of delivering radiation therapy, the two daily doses of MRX 1024 given to patients in cohorts 4 and 5 will be approximately 75 to 90 minutes apart.

To ensure accurate and compliant dosing, MRX-1024 treatment must be administered in the clinic.

Beginning on Day 1 of Week 1 of the Combination Phase, patients will begin receiving MRX 1024 in conjunction with radiation and cisplatin or carboplatin, chemotherapy.

MRX 1024 will be given prior to each day's radiation fraction, and again following each day's radiation fraction for patients being treated in cohorts 4 and 5. If a scheduled radiation treatment is not given, the MRX 1024 dose should not be given on that day.

Dose escalations will occur in successive cohorts as indicated in Table 5 above, based on the rules for dose level escalation as described in Table 6, below. Intra-patient dose escalation is not permitted. No dose adjustments of MRX 1024 are permitted. If a patient experiences a DLT that precludes further treatment with MRX 1024, MRX 1024 treatment will be discontinued. That patient will continue on study, receive radiation therapy and cisplatin or carboplatin, according to the protocol, and be followed on study through the Follow Up Phase.

The next higher dose level will be opened for enrollment after:

1. the preceding dose level has enrolled three patients,
2. two of these patients have completed Days 1 through 42
3. the third patient has completed four weeks of the Combination treatment
4. none of these patients experiencing a dose limiting toxicity.

If one patient being treated in an open dose level experiences a DLT during this interval, then 3 more patients must be enrolled and all six patients in that dose level must be followed for a minimum of the 42 day interval described above before a decision can be made regarding further enrollment and escalation to the next higher cohort. If no additional patient experiences a DLT in that cohort, then the next higher cohort will be opened for enrollment.

If greater than 2 patients in a cohort experience a DLT, then that cohort is considered to have exceeded the maximum tolerable dose level. Three additional patients will then be enrolled to the next lower cohort using that treatment schedule The objective of the dose escalation scheme is to identify a safe, tolerable and potentially efficacious dose level using the once daily dosing schedule and a potentially efficacious dose level using the twice daily dosing schedule of MRX-1024 in which less than 1 of 6 patients experiences a DLT.

Dose Level Escalation Rules

Number of Patients in a cohort with DLTa at a Given Dose Level Escalation Dose Rule 0 out of 3. Enter 3 patients at the next higher dose level. If cohort 3 and or cohort 5 are completed with 0 out of 3 patients experiencing a DLT, then enroll 3 additional patients to each respective cohort. greater than 2 Dose escalation will be stopped. This dose will be declared to have exceeded the maximum tolerable dose. Enroll 3 additional patients at the next lower cohort using that MRX 1024 dosing schedule. If this occurs in cohort 1, 25 mg kg will be used as the next lower dose level.

1 out of 3 Enter 3 more patients in this cohort at this dose level. If 0 of these 3 additional patients experience a DLT , then begin enrollment at the next higher cohort. If 1 or more of these 3 additional patients experience a DLT then dose escalation will be stopped. This dose will be declared to have exceeded the maximum tolerable dose. Enroll 3 additional patients at the next lower cohort using that MRX 1024 dosing schedule. If this occurs in cohort 1, use 25 mg kg as the next lower dose level. Less than 1 out of 6 at the highest tolerable dose level

This is generally the Recommended Dose for subsequent clinical trials. a See Section 4.5 for the definition of Dose-Limiting Toxicity

If a patient does not complete the Combination Treatment Phase for any reason related to intolerance of MRX 1024, this will constitute a DLT and the patient will not be replaced in the study. If a patient does not complete the Combination Treatment Phase for any reason unrelated to MRX 1024 and the patient did not experience a DLT, an additional patient will be enrolled in the study. Data from the original patient will remain as part of the study database but that patient's adverse event experience will not be used to evaluate the safety of MRX 1024 at that dose level.

After the study has ended, an additional analysis of the safety data will be performed to evaluate potential alternate dosing schemes. The doses used in the five dose levels described above will be converted on an individual patient basis to approximate fixed doses and also to mg body surface area dosing. Based on the additional analyses, a preferred dosing scheme will be recommended for subsequent clinical trials.

Radiation Therapy

Radiation therapy begins on Day 1 of Week 1 of the Combination Treatment Phase. Radiation therapy will be administered using daily fractions of 2 Gy given Monday through Friday, five consecutive days each week, followed by two days of no therapy. Radiotherapy will continue weekly in this fashion until the total planned radiation dose of 60 to 66 Gy has been delivered over a 6-week period. The toxicology studies of MRX-1024 were conducted exposing animals for a maximum duration of 27 days. Therefore MRX 1024 can be administered only during the first five weeks of radiation therapy . The sixth week of radiation therapy is not accompanied by treatment with MRX 1024 .

Cisplatin or Carboplatin

Cisplatin will be administered intravenously on Day 1 of Week 1, Day 1 of Week 4 , and on Day 1 of Week 7 using a dose of 100 mg per square meter of body-surface area for cisplatin and AUC5 6 for carboplatin. On these days, the preferred sequence of treatments will be MRX 1024 Radiotherapy . This sequence should allow the MRX 1024 doses to be absorbed before the patient potentially develops vomiting from the chemotherapy. See Section 4.6 for guidelines regarding the use of antiemetics in conjunction with cisplatin or carboplatin dosing.

Cisplatin therapy will include pre- and post treatment hydration requirements according to standard practices within the institution. An example of such hydration procedures follows:

Prior to receiving cisplatin, each patient must receive vigorous hydration and diuresis. A suggested regimen is pre-hydration with a 1 liter of D5NS over 2 to 4 hours and mannitol 12.5 g intravenously bolus immediately prior to cisplatin. Then cisplatin 100 mg m2 in 500 ml NS is administered over 1 to 2 hours with an additional 1 to 1.5 liters of fluid given post-hydration. The type, volume, and rate of fluid administration may vary based on the patient's clinical status and ability to handle the hydration requirement.

Carboplatin therapy will also include the pre- and post-treatment hydration. For the regimen that allows for 21 days recovery the AUC 5-6 dose will be used. The carboplatin dose will be administered with 250 mL NS at 5 mg min mL over 30 minutes.

The dose of cisplatin given on Day 1 of Weeks 4 and 7 is to be adjusted based on the parameters shown below. Laboratory tests used to determine the adjusted cisplatin dose are to be obtained within 3 days prior to the scheduled cisplatin dose. For carboplatin, dose adjustments will be based on laboratory test results obtained within 7 days prior to carboplatin dosing.

Absolute neutrophil count less than 1500 µl: Cisplatin should be held if the ANC less than 1500 µl. After the ANC recovers above this value, the cisplatin dose should be adjusted based on the ANC nadir that was achieved following the preceding cisplatin dose, as shown in Table 7. If the ANC has not recovered within 14 days of when the third cisplatin dose is scheduled , the patient should complete the final Follow-Up Visit without receiving the third dose of cisplatin. For carboplatin, the adjustment will be made if the neutrophil count is less than 1300 mm3.

Platelet count less than 100,000 µl: Cisplatin and carboplatin should be held if the platelet count is less than 100,000µl. After the platelet count recovers above this value, the cisplatin dose should be adjusted based on the platelet count nadir that was achieved following the preceding cisplatin dose, as shown in Table 7. If the platelet count has not recovered within 14 days of when the third cisplatin dose is scheduled , the patient should complete the final Follow Up Visit without receiving the third dose of cisplatin.

Cisplatin Dose Adjustment Based on Absolute Neutrophil Count and Platelet Count Nadirs Following the Preceding Cisplatin Dose Nadir percentage of 100 Cisplatin Dose to Give.

Renal Toxicity: Cisplatin will not be given if the serum creatinine is greater than 1.6 mg dL. Reduce the cisplatin dose for transient rises in serum creatinine as shown in Table 8. Adjustments in the carboplatin dose or or delay in administration will occur if the serum creatinine is greater than 2.0 mg dL.

Liver toxicity: An adjustment in dose or delay in administration will occur if the t. bili is greater than 1.5 mg dL.

Cisplatin Dose Adjustment Based on Highest Serum Creatinine Value Obtained Following the Preceding Cisplatin Dose Serum Creatinine Peak (mg dL)percentage of 100 Cisplatin Dose to Give.

In patients whose serum creatinine does not return to less than 1.6 mg dL by the scheduled day of cisplatin treatment , carboplatin will be substituted and continued at 3 week intervals in lieu of cisplatin.

Neurotoxicity: Cisplatin should be discontinued if any of the following signs of neurotoxicity occur following the first dose of cisplatin: Grade 3 hearing loss in the speech frequency range, Grade 3 myopathy, Grade 3 weakness, Grade 3 neuropathy, seizure or paralysis . If in the Investigator's opinion, said adverse events are related solely to cisplatin, they would not qualify as DLTs. If in the Investigator's opinion, said adverse events may possibly be related to co-administration of MRX 1024, they would qualify as DLTs.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proved squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx;
* Status-post surgical resection of primary disease and meeting criteria for post-operative radiotherapy and chemotherapy by evidence of histologic extracapsular nodal extension, or histologic involvement of >2 regional lymph nodes, or mucosal margin of resection with invasive cancer (limited to microscopic detection only);
* Able to begin protocol treatment within 8 weeks of first tumor-related surgery;
* Age >18 years. Because no dosing or adverse event data are currently available on the use of MRX-1024 in combination with radiotherapy and cisplatin or carboplatin, in patients less than 18 years of age, children are excluded from this study, but will be eligible for future pediatric Phase 1 combination studies in appropriate indications when sufficient safety and efficacy data in adults are available.
* Karnofsky Performance Status of >70 (Appendix I);
* Normal organ and marrow function as defined herein, determined by laboratory values obtained within seven days prior to receiving the first dose of protocol treatment:

  * Serum creatinine within institutional limits of normal
  * Creatinine clearance >50
  * Total bilirubin within institutional limits of normal
  * AST(SGOT) and ALT(SGPT) <2.5 times the upper limit of normal for the institution
  * White blood cell count >3500 per cubic millimeter
  * Absolute neutrophil count >1500 per cubic millimeter
  * Platelet count >100,000 per cubic millimeter
* Ability to understand and the willingness to sign an informed consent document in accordance with institutional guidelines.

Exclusion Criteria:

* Gross (visible or palpable) disease left after surgical resection;
* Prior chemotherapy or radiation therapy to the head and neck region;
* Primary site of the lip, nasopharynx or paranasal sinuses;
* Distant metastases;
* Known malabsorption syndrome;
* Pregnancy or breast-feeding. The effects of MRX-1024 on the developing human fetus are unknown at this time. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately;
* Gastrointestinal tract disease or deformity resulting in an inability to take oral or enteral medication or nutrition;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, untreated or new cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
* History of taking any investigational medication within 4 weeks prior to receiving the first dose of protocol treatment.
* Prior malignancy within the previous 5 years, excluding non-melanoma skin cancer and cervical cancer treated with local therapy.
* Known allergy or sensitivity to polysorbate 80 (Tween).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
safe recommended doses and dose regimen for oral MRX-1024 with concurrent chemoradiation.
Identify toxicity profile of oral MRX-1024.
Determine pharmacokinetic parameters of oral MRX-1024.

SECONDARY OUTCOMES:
Possibly show a trend in activity of MRX-1024 in preventing or reducing oral mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Bajaj, M.D., Principal Investigator — Johns Hopkins University